CLINICAL TRIAL: NCT06123897
Title: Establishing a Clinical Database and Biobank for Schizophrenia：A Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Central South University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Nanjing Brain Hospital, Nanjing Medical University (Unknown); Anhui Mental Health Center (Unknown)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Other Study IDs: WU2023cohort
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Cohort Study
MeSH Terms: conditions — Schizophrenia | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with schizophrenia: Inclusion Criteria:
  * 1.Clinical diagnosis of schizophrenia according to ICD-11.
  * 2.Confirmation of the diagnosis of schizophrenia using the SCID-5-RV (DSM-5 Structured Clinical Interview for DSM-5 Disorders - Research Version).
  Exclusion criteria:
  * 1.Clinical diagnosis or SCID-5-RV assessment confirming neurodevelopmental disorders, bipolar and related disorders, substance use disorders (excluding alcohol and tobacco).
  * 2.Presence of severe or acute physical illnesses, including traumatic brain injury, intracranial space-occupying or infectious diseases, acute cardiovascular diseases, acute respiratory system diseases, acute hematological disorders, etc.
  * 3.Presence of clearly defined genetic diseases, including tuberous sclerosis, multiple sclerosis, Kleefstra syndrome, 22q11.2 deletion syndrome, Prader-Willi syndrome, Klinefelter syndrome (47,XXY), etc.
  Interventions: Other: Regular follow-up assessments without intervention.
- Healthy volunteers: * Inclusion Criteria:
    1. Ages 13-60 years old.
    2. Clinical diagnosis not meeting ICD-11 criteria for schizophrenia.
    3. Diagnosis not meeting schizophrenia criteria confirmed using SCID-5-RV (DSM-5 Structured Clinical Interview for DSM-5 Disorders - Research Version).
  * Exclusion criteria are the same as for the schizophrenia patient group.
  Interventions: Other: Cross-sectional assessment

INTERVENTIONS:
Other: Regular follow-up assessments without intervention. — Participants will undergo follow-up for a minimum of one year, with regular clinical data collection at baseline, half a month, 1st month, 3rd months, 6th months, 9th months and 12th months. Baseline assessments will include demographic information, medical history, and previous medication use. For participants on antipsychotics at baseline, the Simpson-Angus Scale for extrapyramidal symptoms(SAS) will also be administered. At baseline and each follow-up, data on current medication, physical examination, anthropometry, ECG, EEG, psychiatric scales (PANSS, CGI, GAF, PSP, SAS, TESS, MMAS-8), the MATRICS Consensus Cognitive Battery, and laboratory tests (blood routine, liver and renal function, lipids, fasting glucose, fasting insulin, HbA1c) will be obtained, alongside fMRI, eye movement, and fNIRS measures. Blood samples will be collected and stored for mechanistic investigations.
  Groups: Individuals with schizophrenia
Other: Cross-sectional assessment — Volunteers will undergo assessments, including SCID scale, SCL-90, Chinese Perceived Stress Scale(CPSS), the Measurement and Treatment Research to Improve Cognition in Schizophrenia(MATRICS) Consensus Cognitive Battery, blood test(blood routine, liver function, renal function, blood lipids, fasting blood glucose, fasting serum insulin, fasting blood glycosylated hemoglobin), as well as functional MRI, eye movement, functional near-infrared spectroscope and electroencephalogram. Blood samples for exploring difference between patients and healthy people will be collected and stored.
  Groups: Healthy volunteers

SUMMARY:
This is a multicenter study conducted in collaboration with Central South University, The First Affiliated Hospital of Zhengzhou University, Nanjing Brain Hospital of Nanjing Medical University, and Anhui Mental Health Center. The project intends to employ standardized diagnostic criteria and clinical assessment procedures to establish a comprehensive cohort of patients with schizophrenia, encompassing all age groups and disease stages, with follow-up periods exceeding one year. The goal is to create an internationally high-standard clinical cohort database and biobank for schizophrenia. Through a multidimensional assessment framework, the project aims to further investigate the etiology of schizophrenia, patterns of disease progression, and clinical outcomes. By periodically capturing dynamic information on risk and preventive factors, the project aims to achieve early diagnosis, early treatment, and improved prognosis for patients. Additionally, it seeks to explore potential biomarkers within the realm of precision medicine that can predict treatment efficacy, providing viable tools for precision healthcare and clinical decision-making in the field of schizophrenia.

DETAILED DESCRIPTION:
Participants screened through inclusion and exclusion criteria will be recruited and will undergo follow-up for a minimum of one year, with regular clinical data collection at baseline, half a month, 1st month, 3rd month, 6th month, 9th month, and 12th month.The information of demographic data, medical history and previous medication regimen will be collected at baseline. Current medication regimen, physical examination, anthropometry, electrocardiogram, electroencephalogram, psychiatry scales(Positive And Negative Syndrome Scale, Clinical Global Impression, Global Assessment Function and Personal and Social Performance Scale), the Measurement and Treatment Research to Improve Cognition in Schizophrenia(MATRICS) Consensus Cognitive Battery and blood test(blood routine, liver function, renal function, blood lipids, fasting blood glucose, fasting serum insulin, fasting blood glycosylated hemoglobin) will be performed at every follow-up timepoint, as well as functional MRI, eye movement and functional near-infrared spectroscope. If antipsychotic medication is already being used at baseline, the Simpson-Angus Scale (SAS), the Treatment Emergent Symptom Scale (TESS), and the Morisky Medication Adherence Scale (MMAS-8) are administered. Blood samples for exploring underlying mechanisms will be collected and stored at the same time for blood tests.

Data quality control is a crucial step in ensuring the quality and credibility of research data. This project has established a rigorous data quality control system to ensure the rigor and effectiveness of its research work:

1. Establishing management specifications and systems for raw data. Emphasis is placed on protecting the authenticity, integrity, and traceability of raw data, and arbitrary changes are not allowed. In the process of data processing, if there are errors, omissions, or modifications needed, it should follow certain procedures and rules for revision (such as documenting all changes, including detailed information such as time, reasons, values before and after modification, and retaining the original erroneous data as a backup). Trace the entire data processing process to ensure that any changes have clear reasons and evidence support, avoiding the risk of tampering or false reporting.
2. Conduct regular consistency training. This project conducts consistency training for team members on scales and MCCB once every three months, including theoretical explanations, practical operation demonstrations, and practice discussions in various forms. This ensures that all scale assessors understand the design principles, applicability, assessment methods, and scoring criteria of the above scales, thereby reducing errors caused by improper operation.
3. Random inspections. This project also invites senior clinical physicians and researchers to conduct quality control of scale assessments and data collection processes through random inspections. This includes, but is not limited to, reviewing the operating procedures of participating researchers, data recording forms, equipment usage, and other aspects to ensure that all links are within a controllable range and comply with predetermined standards. If any problems or deviations are found, they should be corrected and relevant operating procedures adjusted in a timely manner to ensure continuous improvement in data quality, thereby reducing the error rate and the proportion of invalid data.

ELIGIBILITY:
Inclusion Criteria:

* 1.Clinical diagnosis of schizophrenia according to ICD-11.
* 2.Confirmation of the diagnosis of schizophrenia using the SCID-5-RV (DSM-5 Structured Clinical Interview for DSM-5 Disorders - Research Version).

Exclusion criteria:

* 1.Clinical diagnosis or SCID-5-RV assessment confirming neurodevelopmental disorders, bipolar and related disorders, substance use disorders (excluding alcohol and tobacco).
* 2.Presence of severe or acute physical illnesses, including traumatic brain injury, intracranial space-occupying or infectious diseases, acute cardiovascular diseases, acute respiratory system diseases, acute hematological disorders, etc.
* 3.Presence of clearly defined genetic diseases, including tuberous sclerosis, multiple sclerosis, Kleefstra syndrome, 22q11.2 deletion syndrome, Prader-Willi syndrome, Klinefelter syndrome (47,XXY), etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from outpatient or inpatient departments.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the MATRICS Consensus Cognitive Battery score | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  After assessment at each visit, evaluator convert raw scores to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated. The changes of scores at different follow up timepoint will be used for assessing the improvement of cognitive function (higher score means a better outcome).
Change of clinical symptoms by Positive And Negative Syndrome Scale | baseline, half a month, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  The change of Positive And Negative Syndrome Scale at different follow up timepoint (lower score means a better outcome)
Change of clinical symptoms by Clinical Global Impression | baseline, half a month, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  The change of Clinical Global Impression at different follow up timepoint (lower score means a better outcome)

SECONDARY OUTCOMES:
Change of the level of blood lipids | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Blood lipids include total cholesterol, low-density lipoprotein-cholesterol, triglyceride and high-density lipoprotein-cholesterol.
Change of Body Mass Index | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  BMI = weight/height^2,To some extent, Body Mass Index(BMI) can represent the situation of peripheral metabolism.
Change of waist-hip circumference | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Change of waist-hip circumference,To some extent, waist-hip circumference can represent the situation of peripheral metabolism.
Changes of the level of fasting blood glucose | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Changes of fasting blood glucose
Changes of the level of fasting insulin | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Changes of fasting insulin
Changes of the level of fasting glycated hemoglobin | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Changes of fasting glycated hemoglobin
Changes of functional MRI | baseline, 3rd month, 6th month, 9thmonth, 12th month
  Resting functional MRI will be acquired using a Fast Echo-Planar Imaging (FE-EPI) sequence based on Blood Oxygenation Level Dependent (BOLD) contrast.
Changes of eye movement | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Eye-tracking data will be collected using the EyeLink 1000 eye-tracking system from SR Research. The sampling frequency was 1000 Hz. Stimuli will be presented on a 24-inch computer monitor with a refresh rate of 120 Hz, and the viewing distance will be 70 centimeters. Eye movement data extraction and filtering will be performed using the Data Viewer 3.2 software, which is compatible with the EyeLink system.
Changes of brain hemodynamics detected by functional near-infrared spectroscope system | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Changes of brain hemodynamics detected by functional near-infrared spectroscope system
Change of electroencephalogram | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Neuroscan multi-channel evoked potential workstation records EEG data, using the international 10-20 system for electrode placement, with Ag/AgCl electrodes on a 64/128 electrode cap.
Change of social function by Personal and Social Performance Scale | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Change of social function by Personal and Social Performance Scale, higher score means a better outcome.
Change of Global Assessment Function | baseline, 1st month, 3rd month, 6th month, 9thmonth, 12th month
  Change of Global Assessment Function (GAF), higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, M.D., Ph.D., Study Chair — Mental Health Institute of Second Xiangya Hospital,CSU
Locations (4):
- China (4):
  - Anhui Mental Health Center, Hefei, Anhui
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Mental Health Institute of Second Xiangya Hospital,CSU, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuan H, Wang MY, Liu RX, Sreekissoon S, Liu Q, Tan L, Zhao YQ, Zhong MM, Zhang Q, Su XL, Chen NX, Wang M, Yang YF, Li JN, Zheng HQ, Chen JD, Feng YZ, Zhang FY, Guo Y. Olanzapine affects bone formation via oral Enterococcus through SAA1 gene and extracellular matrix-related pathways. Front Cell Infect Microbiol. 2026 Jan 6;15:1673931. doi: 10.3389/fcimb.2025.1673931. eCollection 2025. PMID 41568002